CLINICAL TRIAL: NCT06636058
Title: Digital InteGrated Behavioral TreatmeNt for Comorbid ObesITy and DeprEssion Among Racial and Ethnic Adults Age 50 and Older (IGNITE)
Brief Title: Digital InteGrated Behavioral TreatmeNt for Comorbid ObesITy and DeprEssion Among Racial and Ethnic Adults Age 50 and Older
Acronym: IGNITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Washington University School of Medicine (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Principal Investigator, Beth and George Vitoux Professor of Medicine Affiliation: University of Illinois at Chicago, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0908; R01AG084527 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Depression
MeSH Terms: conditions — Obesity; Depression | interventions — Maintenance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early VCare Intervention (6-month active treatment followed by 6-month maintenance) (Experimental): Participants randomized to the early-intervention arm will receive active treatment for 6 months, followed by maintenance for another 6 months.
  Interventions: Behavioral: vCare Intervention (6-month active treatment followed by 6-month maintenance)
- Later Waitlist VCare Intervention (active treatment after 6 months) (Active Comparator): Participants in the later-intervention arm will be waitlisted for 6 months and then receive active treatment in the second 6 months.
  Interventions: Behavioral: vCare Intervention (active treatment after 6 months)

INTERVENTIONS:
Behavioral: vCare Intervention (6-month active treatment followed by 6-month maintenance) — During the active treatment, participants will interact with the Lumen virtual coach (for depression management) and watch the GLB videos (for weight loss). Using the Amazon Alexa app on their study iPads, participants will complete 4 weekly Lumen PST sessions initially, 2 bi-weekly sessions, and then 3 monthly sessions during the active intervention. Beginning in week 6, participants will receive automated messages with instructions to view one GLB video a week for 11 weeks.
  During the maintenance period, participants in the early vCare intervention arm will be able to interact with Lumen for PST coaching when they need to, i.e., "on demand," although they will receive reminders to do so at least once a month. Participants may watch any of the 12 GLB videos again and will receive GLB-themed reinforcement and motivational messages by email every 2 weeks.
  Arms: Early VCare Intervention (6-month active treatment followed by 6-month maintenance)
Behavioral: vCare Intervention (active treatment after 6 months) — During the active treatment, participants will interact with the Lumen virtual coach (for depression management) and watch the GLB videos (for weight loss). Using the Amazon Alexa app on their study iPads, participants will complete 4 weekly Lumen PST sessions initially, 2 bi-weekly sessions, and then 3 monthly sessions during the active intervention. Beginning in week 6, participants will receive automated messages with instructions to view one GLB video a week for 11 weeks.
  Arms: Later Waitlist VCare Intervention (active treatment after 6 months)

SUMMARY:
The goal of this randomized clinical trial is to test the efficacy of a fully digital intervention, combining the Lumen problem-solving therapy virtual coach for depression management with the Diabetes Prevention Program video-based program for weight loss, among racial and ethnic minorities with comorbid depression and obesity. The study aims include:

* Determine the efficacy of the vCare intervention at 6 months. Primary outcomes are weight and depression symptom checklist 20-item (SCL-20) score.
* Identify predictors of treatment success, defined by achieving clinically significant weight loss (5%) and depression outcomes (50% decline or SCL-20<0.5), at 6 and 12 months.
* Characterize participant experiences and perceptions of the vCare intervention. Eligible participants will be randomized to the early-intervention arm who will receive active treatment for 6 months, followed by maintenance for another 6 months, or the later-intervention arm who will be waitlisted for 6 months and then receive active treatment in the second 6 months.

DETAILED DESCRIPTION:
The objective of this project is to test the efficacy of a fully digital intervention, combining the Lumen problem-solving treatment (PST) virtual coach for depression management with the Diabetes Prevention Program (DPP) video-based program for weight loss. This integrated intervention is named vCare. Patients self-identified as a racial or ethnic minority with depression and obesity will be enrolled from a large minority-serving academic medical center in Chicago.

In this fully remote clinical trial, participants will receive a study iPad, a wireless weight scale, and a wearable activity tracker. Eligible participants who complete baseline assessment (N=440) will be randomly assigned in 1:1 ratio to receive the vCare intervention early (for 6 months of active treatment and 6 months of maintenance) or later (for 6 months waitlist control and 6 months of active treatment). Participants in either the early- or later-intervention arm will be assessed at 6 and 12 months follow-up.

The specific aims of this study are to (1) determine the intervention efficacy to improve the primary depressive symptoms and weight loss outcomes and secondary outcomes (e.g., anxiety, sleep, quality of life, social isolation, loneliness, and psychosocial and cognitive functioning) at 6 months; (2) identify predictors of treatment success, defined by clinically significant weight loss (5%) and depression response (50% symptom reduction) or remission (free of symptoms), at 6 and 12 months; and (3) characterize the experiences and perceptions of intervention participants to inform future adaptation and translation.

ELIGIBILITY:
Inclusion Criteria

* Age 50-74 years (inclusive)
* Confirmed body mass index (BMI) between ≥27.0 and <45.0 based on weight and height measured by study staff at device distribution
* Confirmed weight ≤396 lbs
* Patient Health Questionnaire-9 (PHQ-9) scores between ≥10 and <20, indicating moderate to moderately severe depressive symptoms
* Self-identified race and ethnicity other than non-Hispanic White
* Willing and able to accept randomization, and provide informed e-consent and HIPAA authorization

Exclusion Criteria

* Unable to speak, read, understand English sufficiently for informed consent
* No reliable Wi-Fi Internet access at home
* Pre-existing type 1 or type 2 diabetes, coronary heart disease, heart failure, stroke, cancer diagnosis (other than non-melanoma skin cancer) or treatment in the past 12 months, end-stage organ failure, residence in a long-term care facility, life expectancy <24 months
* Self-report of weight change >15 lbs. during prior 3 months
* Current active weight loss treatment, including research-based commercial weight loss programs (e.g., Weight Watchers, Jenny Craig, HMR, Omada, TOPS), other programs led by trained personnel (professional or lay) at the recruiting clinic or in the local community
* Taking prescription medications regularly that affect appetite/weight (e.g., anti-obesity medicines, oral corticosteroids, oral hypoglycemics, etc.) for chronic disease management
* Planned or prior bariatric surgery (Note: patients who are more than 2 years post bariatric surgery may otherwise be eligible)
* Screen positive for bulimia nervosa using PHQ- eating disorder module
* Unable to pass the Revised Physical Activity Readiness Questionnaire (PAR-Q) or obtain physician clearance to participate
* Active suicidal ideation (PHQ-9 item 9 score ≥1 or SCL-20 item 2 score ≥2) with active plan and/or intent
* Bipolar or psychotic disorder, or pharmacotherapy or psychotherapy (individual or professionally-led group therapy), or brain stimulation therapy for depression or any other psychiatric condition
* Cognitive impairment based on the Callahan 6-item screener
* Active alcohol or substance use disorder (including prescription drugs) based on the CAGE Questionnaire Adapted to Include Drugs (CAGE-AID)
* Current or planned pregnancy or lactating (<6 months postpartum)
* Participation in other behavioral, medical or surgical treatment studies by self-report that conflict with the primary weight loss and depression outcomes of this study
* Family/household member of an already enrolled participant or of a study team member
* Investigator discretion for serious safety or protocol adherence reasons

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-04-14 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Changes in weight from baseline to 6 months | From Baseline to 6 months
  All participants will receive a study-provided wireless weight scale (Withings Body - Digital Wi-Fi Smart Scale), assistance with account and device setup, and as-needed tech support. A study coordinator who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to weigh themselves in the morning after urination (and a bowel movement too, if able to do so) on 3 days during the assessment week at baseline (0), 6, 12 months. Participants will be instructed to self-weigh in a T-shirt and undergarment and with no socks or shoes using their study-provided digital scale. We will obtain participants' self-monitored weight data using a developed program for automated daily synchronization via the Fitbit open API.
Changes in Depression Symptom Checklist 20-items (SCL-20) from baseline to 6 months | From Baseline to 6 months
  The SCL-20 is a valid, reliable measure of depression severity. It has been used in numerous depression treatment trials in primary care and community settings, making it particularly useful for cross-study comparisons and data synthesis in meta-analyses. The SCL-20 had good internal consistency (Cronbach's alpha=0.859) and correlated well with the General Health Questionnaire (r=0.78), a psychiatric screening test.

SECONDARY OUTCOMES:
Changes in weight from baseline to 12 months | From Baseline to 12 months
  All participants will receive a study-provided wireless weight scale (Withings Body - Digital Wi-Fi Smart Scale), assistance with account and device setup, and as-needed tech support. A study coordinator who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to weigh themselves in the morning after urination (and a bowel movement too, if able to do so) on 3 days during the assessment week at baseline (0), 6, 12 months. Participants will be instructed to self-weigh in a T-shirt and undergarment and with no socks or shoes using their study-provided digital scale. We will obtain participants' self-monitored weight data using a developed program for automated daily synchronization via the Fitbit open API.
Changes in Depression Symptom Checklist 20-items (SCL-20) from baseline to 12 months | From Baseline to 12 months
  The SCL-20 is a valid, reliable measure of depression severity. It has been used in numerous depression treatment trials in primary care and community settings, making it particularly useful for cross-study comparisons and data synthesis in meta-analyses. The SCL-20 had good internal consistency (Cronbach's alpha=0.859) and correlated well with the General Health Questionnaire (r=0.78), a psychiatric screening test.
Clinically significant weight change from baseline | From baseline to 6 months, 12 months
  Dichotomous variable based on if participants reaching 5% weight loss from baseline.
Depression Response | From baseline to 6 months, 12 months
  Dichotomous variable based on if participants achieving 50% decline in Depression Symptom Checklist (SCL-20) scores from baseline.
Depression Remission | Baseline, 6 months, 12 months
  Dichotomous variable based on if participants achieving Depression Symptom Checklist (SCL-20) scores <0.5.
Changes in Generalized Anxiety Disorder 7-item (GAD-7) from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Anxiety will be measured with the Generalized Anxiety Disorder Scale (GAD-7). GAD-7 is a valid and reliable 7-question scale for screening generalized anxiety disorder and strongly associated with multiple domains of functional impairment. It has excellent internal consistency (Cronbach's alpha=0.92) and good test-retest reliability (intraclass correlation=0.83). GAD-7 correlated well with the Beck Anxiety Inventory (r=0.72) and the anxiety subscale of the Symptom Checklist-90 (r=0.74).
Changes in Sleep disturbance and impairment from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Sleep disturbance will be assessed on the 8-item PROMIS sleep disturbance (SD) scale. SD measures symptoms of insomnia. Each item is scaled from 1 (not at all) to 5 (very much). Correlation between the SD short form and the Pittsburgh Sleep Quality Index (PSQI, hypothesized to measure similar attributes) is 0.83, similar to the correlations between the SD full banks and PSQI (0.85).
Changes in Sleep impairment from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Sleep impairment will be assessed on the 8-item PROMIS sleep-related impairment (SRI) scale. SRI measures symptoms of daytime sleepiness. Each item is scaled from 1 (not at all) to 5 (very much). Correlation between the SRI short form and the Epworth Sleepiness Scale (ESS, hypothesized to measure a related but slightly different construct, the propensity to doze during activities) is 0.46, similar to the correlations between SRI full banks and the ESS (0.45).
Changes in functional impairment from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  The Work and Social Adjustment Scale (WSAS) is a validated questionnaire that measures impaired functioning. Patients rate the extent to which their depression symptoms impair work, home management, leisure activities, and relationships with others on a 0 (no impairment at all) to 8 (very severe impairment) scale. Cronbach's alpha ranged from 0.70-0.94. Test-retest correlation was 0.73.
Changes in Cognitive functioning from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  The PROMIS Cognitive Abilities and Cognitive Concerns Scales each contain 8 items. The Cognitive Abilities items positively worded and the Cognitive Concerns items are worded negatively. Items on both subscales use a 5-point rating from "not at all" to "very much." Items are summed to create a total score for each subscale. Cronbach's α coefficients were 0.94 for both scales. The test-retest correlation coefficients were 0.83 for Cognitive Concerns and 0.80 for Cognitive Abilities over a 2-month period. A total score was calculated by summing item scores with reverse coding the Concerns subscale items. Higher total scores indicate better cognitive function.
Changes in Obesity-related quality of life from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  The Obesity-Related Problem Scale specifically measures the impact of obesity on psychosocial functioning. The 8-item scale has internal reliability (Cronbach's a) above 0.90. The scale correlates strongly with theoretically related constructs and weight loss. The scale among the obese was significantly related to poor mood measured with the Mood Adjective Check List (MACL) (P<0.0001) and anxiety and depression symptoms measured with the Hospital Anxiety and Depression Scale (HAD) (P<0.0001). Change in scale over time was strongly correlated with weight loss (P<0.0001).
Changes in Generic health-related quality of life from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  The 8-item Short-Form Health Survey (SF-8) is an 8-item version of the SF-36 that measures overall health-related quality of life. Physical and mental health composite scores are computed using the scores of 8 questions and range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health. Correlation between the SF-8 and the SF-36 is 0.825 for physical health component and 0.881 for mental health component.
Changes in Social isolation from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Social Network Index measures ties in four domains: marriage or partnership, friends and relatives, religious activity, and voluntary associations. Scores for the four dichotomized variables are summed with a range of 0 to 4, with a score of 4 indicating social ties across all four domains. Each type of social die significantly associated with lower mortality rate, independent of the other three.
Changes in loneliness from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Loneliness will be measured with the UCLA 3-item Loneliness Scale, with response categories being 1 (hardly ever), 2 (some of the time), and 3 (often). Responses to the 3 questions are summed, with higher scores representing greater loneliness. The Cronbach's alpha is 0.72. The 3-item loneliness scale significantly correlated with the 20-item Revised UCLA Loneliness Scale (r=0.82), depressive symptoms measured by a short form of the Center for Epidemiologic Studies-Depression Scale (CES-D) (r=0.48-0.49), and the 4-item Perceived Stress Scale (r=0.40-0.44).
Changes in physical activity from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  All participants will receive a study-provided Fitbit activity tracker with heart rate and sleep monitor, assistance with account and device setup, and as-needed tech support. A study coordinator who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to wear their activity tracker for at least 10 hours on 3 or more days during the assessment week at baseline (0), 6, 12 months. We will obtain participants' self-monitored activity and heart rate data using a developed program for automated daily synchronization via the Fitbit open API.
Changes in sleep metrics from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Sleep data will be obtained from Fitbit Alta HR activity trackers following the same procedures as described above for physical activity assessment at 0, 6, and 12 months.
Changes in diet intake from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Dietary intake will be measured using 17-item fruit, vegetable, fat, and fiber screener by self-report. Correlations between screener estimates and estimated true intake were 0.5-0.8.
Changes in problem-solving ability from baseline to 6, 12 months | From Baseline to 6 months, 12 months
  Social Problem-Solving Inventory-Revised: Short Form (SPSI-R:S) assesses participants' problem-solving abilities. The scale is reliable and valid, containing 25 items in the following 5 subscales: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving (RPS), impulsive/careless style (ICS), and avoidance style (AS). Each item is rated on a 5-point scale ranging from "not at all true of me" (0) to "extremely true of me" (4). SPSI-R:S is a short version of the long SPSI-R:L form which has Cronbach's alpha coefficient of 0.95 for the total score and of 0.67-0.92 for subscales.
Changes in food insecurity from baseline to 12 months | From Baseline to 12 months
  Food insecurity will be measured with the 2-item Seattle Short form at baseline and 12 months. The 2 questions are about the food eaten in your household in the LAST 12 MONTHS, and whether you were able to buy the food you needed. Compared with the 6-item screen, the 2-item screen was found to have 95.4% sensitivity and 83.5% specificity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Department of Medicine, Vitoux Program on Aging and Prevention, Chicago, Illinois
  - Washington University School of Medicine in St Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided
IPD under development